CLINICAL TRIAL: NCT00557557
Title: A Phase I Trial of Isolated Hepatic Perfusion With Oxaliplatin and 5-fluorouracil (5-FU) Followed by Hepatic Arterial Infusion of FUDR for Patients With Unresectable Colorectal Liver Metastases
Brief Title: Safety Study of Oxaliplatin and 5-fluorouracil Followed by FUDR for Unresectable Colorectal Liver Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: David Bartlett (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, David Bartlett, Chief, Division of Surgical Oncology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-096; 1R21CA115059-01A1 (NIH)
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-12

CONDITIONS: Colorectal Liver Metastases
Keywords: Colorectal; liver; cancer; metastases
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — Fluorouracil; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IHP with Oxaliplatin and 5-Fluorouracil (5-FU) (Experimental): Isolated Hepatic Perfusion with Oxaliplatin and 5-Fluorouracil (5-FU)
  Interventions: Drug: Drug: 5-FU; Drug: Drug: Oxaliplatin

INTERVENTIONS:
Drug: Drug: 5-FU — Dose escalation (200 to 900 mg/m²) scheme, one hour isolated hepatic perfusion prior to standard treatment.
Drug: Drug: Oxaliplatin — 40 mg/m², one hour isolated hepatic perfusion prior to standard treatment.

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose and dose limiting toxicity of 5-FU in combination with Oxaliplatin delivered via isolated hepatic perfusion.

DETAILED DESCRIPTION:
Subjects who are planning to undergo surgery for placement of HAI therapy pump will be considered for enrollment. Standard HAI therapy requires a laparotomy and placement of an intrahepatic arterial catheter that is connected to one of several commercially available subcutaneous electronic pumps. The pump is then used to deliver FUDR directly to the liver, usually beginning four weeks after surgery and lasts on average for a period of six to twelve months after the study. Current HAI therapy regimens often alternate FUDR with systemic chemotherapy. This study will examine the addition of a one hour isolated hepatic perfusion with 5-FU and Oxaliplatin prior to this standard treatment. Subjects will be given the consent form to review and after sufficient time to review the information, interested subjects will have the opportunity to ask questions of the investigators. Subjects interested in enrolling in the trial will then sign informed consent and clinical data will be collected from their chart to ensure that they meet eligibility requirements. The study will consist of a one hour isolated liver perfusion that will be performed at the time of the laparotomy to place the HAI therapy pump. Following surgery subjects will be monitored in the ICU for 24-48 hours and potentially in the hospital for an additional 5-7 days. Subjects will be free to start standard HAI therapy regimens four to six weeks following surgery. The duration of treatment, dose of HAI therapy and the decision to combine HAI with systemic chemotherapy will be at the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven measurable metastatic colorectal cancer limited to the parenchyma of the liver by preoperative radiological studies. Limited resectable extrahepatic disease is acceptable if the liver is felt to be the dominate site of life threatening disease.
* No chemotherapy, radiotherapy, or biologic therapy for their malignancy in the 4 weeks prior to the liver perfusion and must have recovered from all side effects.
* An ECOG performance standard of 0, 1 or 2 for 24 hours prior to surgery.
* Adequate hepatic function as evidenced by bilirubin < 2.0 mg/dL and a PT < 2 seconds greater than the upper limit of normal.
* Age equal to 18 years or older and greater than 30 kg.
* Platelet counts greater than 100,000, a hematocrit > 27.0, a white blood count > 3000/µl, Absolute neutrophil count > 1,500/μL and a creatinine less than or equal to 1.5 mg/dL or a creatinine clearance of > 60 mL/min. Patients with elevations in hepatic transaminases secondary to the presence of metastatic disease in the liver are eligible.
* Adequate hepatic function as evidenced by:

  * Serum total bilirubin < 1.5 mg/dL
  * Alkaline phosphatase < 5X the ULN
  * SGOT/SGPT < 5X the ULN
* Aware of the neoplastic nature of his/her illness, the experimental nature of the therapy, alternative treatments, potential benefits, and risks and willing to sign an informed consent.
* The disease in the liver must be considered unresectable as defined by greater than three sites of disease in the liver, bilobar disease, and tumor abutting major vascular or ductal structures making anatomic resection with preservation of liver function impossible.
* Patients of childbearing potential and their partners must agree to use an effective form of contraception during the study and for 90 days following the last dose of study medication

Exclusion Criteria:

* Pregnant patients and nursing mothers will be excluded due to the unknown effects of oxaliplatin on the fetus or newborn.
* Patients with active CNS metastases. Patients with stable CNS disease, who have undergone radiotherapy at least 4 weeks prior to the planned first protocol treatment and who have been on a stable dose of corticosteroids for >3 weeks are eligible for the trial.
* Patients taking immunosuppressive drugs or on chronic anticoagulation will not be eligible.
* Patients with active infections or with a fever > 101.30 F within 3 days of the first scheduled day of protocol treatment are not eligible.
* Patients with biopsy proven cirrhosis or evidence of significant portal hypertension manifested by ascites, esophageal varices on endoscopy, or radiologic studies showing significant collateral vessels around the organs drained by the portal venous system will be excluded.
* Patients with ischemic cardiac disease or history of congestive heart failure with an LVEF < 40% will be excluded.
* Patients with COPD or other chronic pulmonary disease with PFTs indicating an FEV< 50% predicted for age will be excluded.
* Patients with a history of veno-occlusive disease of the liver are ineligible.
* History of prior malignancy within the past 5 years except for curatively treated basal cell carcinoma of the skin, cervical intra-epithelial neoplasia, or localized prostate cancer with a current PSA of < 1.0 mg/dL on 2 successive evaluations, at least 3 months apart, with the most recent evaluation no more than 4 weeks prior to entry.
* Patients with known hypersensitivity to any of the components of oxaliplatin (or combination drug, if any).
* Patients who received radiotherapy to more than 25% of their bone marrow; or patients who received any radiotherapy within 4 weeks of entry.
* Patients who are receiving concurrent investigational therapy or who have received investigational therapy within 30 days of the first scheduled day of protocol treatment (investigational therapy is defined as treatment for which there is currently no regulatory authority approved indication).
* Peripheral neuropathy ≥ Grade 2.
* Any other medical condition, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results.
* History of allogeneic transplant.
* Known HIV or Hepatitis B or C (active, previously treated or both).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-07; Primary Completion 2012-03 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Primary endpoint is to determine the maximum tolerated dose and dose limiting toxicity of 5-FU delivered with 40mg/m² of Oxaliplatin via IHP. | 24 to 48 hours

SECONDARY OUTCOMES:
Secondary endpoints will be to determine the response rate and survival after IHP with 5-FU and Oxaliplatin. | 3 to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Herbert J. Zeh, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Cancer Centers Network, Pittsburgh, Pennsylvania, United States